CLINICAL TRIAL: NCT05614453
Title: A Phase II Trial of Tislelizumab in Combination With Sitravatinib for Recurrent/Metastatic Cervical Cancer After Platinum-Based Chemotherapy
Brief Title: Tislelizumab in Combination With Sitravatinib for Recurrent/Metastatic Cervical Cancer After Platinum-Based Chemotherapy
Acronym: ITTACC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: BeiGene has withdrawn their support owing to sitravatinib supply concerns. Mirati is ceasing further development of sitravatinib owing to the negative results of the SAPPHIRE trial which used sitravatinib in 2nd line met NSCLC setting.
Sponsor: Australia New Zealand Gynaecological Oncology Group (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANZGOG 2002/2021
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tislelizumab; sitravatinib

STUDY DESIGN:
Intervention Model Description: Phase II, open-label, multi-centre study, based on Simon's two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Tislelizumab 200mg (IV) every 21 days for up to 35 cycles Sitravatinib 100mg (oral) given daily until disease progression or unacceptable toxicity
  Interventions: Drug: Tislelizumab; Drug: Sitravatinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab is an investigational, humanised-IgG4 monoclonal antibody with high affinity/binding specificity for PD-1. It is engineered to minimise binding to FcγR on macrophages to abrogate antibody-dependent cellular phagocytosis.
  Other Names: BGB-A317
Drug: Sitravatinib — Sitravatinib is an orally bioavailable receptor tyrosine kinase (RTK) inhibitor with potential anti-neoplastic activity.
  Other Names: MGCD516

SUMMARY:
The goal of this clinical trial is to learn about the effect of the combination treatment of sitravatinib with tislelizumab in patients with Recurrent/Metastatic Cervical Cancer after Platinum-Based Chemotherapy.

The main question it aims to answer is the percentage of people in the study who have a partial or complete response to the treatment.

Participants will receive treatment under the care of their treating physician and will be reviewed regularly.

DETAILED DESCRIPTION:
Monoclonal antibodies that target either PD-1, PD-L1, or the other checkpoint inhibitors can block binding and boost the immune response against cancer cells. However, many early-phase studies with single immune checkpoint inhibitors did not show enough power to achieve a promising clinical response, and several trials are evaluating different strategies to overcome immune tolerance via combination therapies. Combining an immunotherapeutic PD-1 checkpoint inhibitor with an agent that has both immune modulatory and antitumor properties could enhance the antitumor efficacy observed with either agent alone.

Sitravatinib is a spectrum selective RTK inhibitor that inhibits several closely related RTKs, including the TAM family (Tyro3/Axl/MER), VEGFR2, KIT, and MET. Tislelizumab is a humanised IgG4-variant monoclonal antibody against PD-1. In addition to the antiangiogenesis activity of sitravatinib, sitravatinib in combination with tislelizumab may elicit greater anti-tumour activity, as sitravatinib is predicted to enhance several steps in the cancer immunity cycle that may augment the efficacy of tislelizumab.

In summary, sitravatinib inhibits key molecular and cellular pathways strongly implicated in carcinogenesis and drug resistance and represents a reasonable strategy to enhance anti-tumour immunity when combined with tislelizumab.

The ITTACc study aims to assess the overall response rate of the combination of tislelizumab with sitravatinib along with other key outcomes detailed below.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Patient must be ≥ 18 years of age at screening
3. Recurrent, persistent, and/or metastatic cervical cancer with squamous cell histology, adeno-squamous carcinoma, and adenocarcinoma for which there is not a curative-intent option (surgery or radiation therapy with or without chemotherapy)
4. Measurable disease, as defined by RECIST 1.1
5. ECOG performance status ≤ 2
6. Adequate bone marrow, hepatic and renal function documented within 10 days prior to registration, defined as:

   * Haemoglobin ≥ 90g/L
   * ANC ≥ 1.5 x 109/L
   * Platelets ≥ 75 x 109/L
   * Total bilirubin ≤ 1.5x ULN if liver metastases ≤ 3x ULN. Patients with Gilbert's syndrome, and total bilirubin up to 3x ULN may be eligible after communication with and approval from the CPI
   * AST and ALT ≤ 3x ULN (or ≤ 5.0x ULN, if liver metastases)
   * ALP ≤ 2.5x ULN (or ≤ 5.0x ULN, if liver or bone metastases)
   * Serum creatinine ≤ 1.5x ULN or estimated creatinine clearance > 45mL/min using the Cockcroft-Gault equation
7. Patients must meet at least one of the following criteria regarding prior bevacizumab therapy:

   * Received prior bevacizumab-containing therapy, which was discontinued due to progression of disease
   * Received prior bevacizumab-containing therapy, which was discontinued due to toxicity
   * Was deemed unsuitable for prior bevacizumab therapy for one of the following reasons: (i) unacceptable risk of fistula formation, (ii) poorly controlled hypertension, (iii) "low risk" disease according to the Moore Criteria
   * Refused prior bevacizumab therapy
8. Patients must meet at least one of the following criteria regarding prior paclitaxel therapy:

   * Received prior paclitaxel-containing therapy, which was discontinued due to progression of disease
   * Received prior paclitaxel-containing therapy, which was discontinued due to toxicity
   * Was deemed unsuitable for prior paclitaxel therapy for one of the following reasons:

     * Significant neuropathy
     * Allergy to paclitaxel or its components
   * Refused prior paclitaxel therapy
9. 1 prior line of combination which include an anti-PD-1/ anti-PD-L1 inhibitor
10. Previous progression after cisplatin or carboplatin-based combinations
11. Anticipated life expectancy > 12 weeks
12. Willing and able to comply with clinic visits and study-related procedures
13. Availability of archival tumour sample from either the primary or metastatic tumour. If no archival tumour is available, a fresh tissue biopsy to be performed if feasible and safe to do so. Where tumour tissue is not available, this will not preclude trial participation

Exclusion Criteria:

1. Ongoing or recent (within 5 years prior to registration) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest higher risk for severe irAEs. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment
2. Prior treatment with other systemic immune-modulating agents that was (a) within fewer than 28 days prior to registration, or (b) associated with irAEs of any grade within 90 days prior to registration, or (c) associated with toxicity that resulted in discontinuation of the immune-modulating agent.
3. Known history of brain metastasis(es) that may be considered active (screening imaging of brain is not required unless there is clinical suspicion of brain metastases). Patients with previously treated brain metastases may participate provided that the lesions are stable (without evidence of progression for at least 6 weeks on imaging obtained during the screening period), there is no evidence of new or enlarging brain metastases, and the patient does not require any immunosuppressive doses of systemic corticosteroids for management of brain metastases within 4 weeks prior to registration
4. Variant histology's such as high-grade neuroendocrine carcinoma, small cell carcinoma, mucinous carcinoma, sarcomatous tumours or mixed histology's containing these components
5. Patients with tumour shown by imaging to be located around important vascular structures or if the Investigator determines that the tumour is likely to invade important blood vessels and may cause fatal bleeding (i.e., radiological evidence of tumours invading or abutting major blood vessels)
6. Any of the following cardiovascular risk factors:

   * Cardiac chest pain, defined as moderate pain that limits instrumental ADL, ≤ 28 days prior to registration
   * Symptomatic pulmonary embolism ≤ 28 days prior to registration
   * Any history of acute myocardial infarction ≤ 6 months prior to registration
   * Any history of heart failure meeting NYHA Classification III or IV ≤ 6 months prior registration
   * Any ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months prior to registration
   * QTc ≥ 470msec in females and ≥ 450msec in males (based on average of screening triplicates)
   * Cardiac LVEF ≤ 50% or lower limit of normal as assessed by echocardiography or MUGA
   * Patients with inadequately controlled hypertension (defined as systolic blood pressure > 150mmHg and/or diastolic blood pressure > 100mmHg, that is persistent)
   * Any history of cerebrovascular accident ≤ 6 months prior to registration
7. Significant bleeding and thrombotic risks:

   * Patients with bleeding or thrombotic disorders or who use anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring
   * Patients with signs or history of significant bleeding, within 4 weeks prior to registration, patients with any bleeding events ≥ CTCAE Grade 3, unhealed wounds, ulcers, or fractures
   * Patients with arterial thrombotic event that occurred within 6 months prior to
   * registration, such as cerebrovascular accident (including temporary ischemic attack)
   * Venous thrombotic events such as deep vein thrombosis and pulmonary embolism that causes haemodynamic compromise or venous thrombotic events within 4 weeks of diagnosis (treated asymptomatic patients > 4 weeks after diagnosis permitted at Investigators' discretion)
8. Immunosuppressive corticosteroid doses (> 10mg prednisone daily or equivalent) within 4 weeks prior to registration
9. Active bacterial, viral, fungal or mycobacterial infection requiring therapy, including known infection with HIV, or active infection with HBV or HCV
10. History of pneumonitis within the last 5 years
11. Any anticancer treatment (chemotherapy, targeted systemic therapy, photodynamic therapy), investigational, or standard of care, within 30 days prior to registration or planned to occur during the study period (patients receiving bisphosphonates or denosumab are not excluded)
12. History of documented allergic reactions or acute hypersensitivity reactions attributed to antibody treatments
13. Concurrent malignancy other than cervical cancer and/or history of malignancy other than cervical cancer within 3 years prior to registration, except for tumours with negligible risk of metastasis or death, such as adequately treated cutaneous squamous cell carcinoma or basal cell carcinoma of the skin or ductal carcinoma in situ of the breast. Patients with hematologic malignancies (e.g., CLL) are excluded
14. Any acute or chronic psychiatric problems that, in the opinion of the Investigator, make the patient ineligible for participation
15. Patients with a history of solid organ transplant (patients with prior corneal transplant(s) may be allowed to enrol after discussion with and approval from the CPI)
16. Any medical co-morbidity, physical examination finding, or metabolic dysfunction, or clinical laboratory abnormality that, in the opinion of the Investigator, renders the patient unsuitable for participation due to excessive safety risks and/or potential to affect interpretation of results of the study
17. Pregnant or breastfeeding persons
18. People of Childbearing Potential who are unwilling to practice highly effective contraception prior to the initial study drug treatment, during the study, and for at least 6 months after the last dose.
19. Prior treatment with idelalisib
20. Prior treatment with live vaccines within 30 days prior to registration. Patients must not be treated with live vaccines during the study and up to 5 half-lives following the last dose of study drug
21. Patients with prior treatment on any clinical trial within 30 days prior to registration. Non-interventional and observational trials are acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years
  To assess the ORR of the combination of tislelizumab with sitravatinib using RECIST 1.1

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  To estimate OS at 12 months. Defined as the time from the start of treatment until death of any cause.
Progression Free Survival (PFS) | Up to 4 years
  To determine PFS, defined as the time from start of treatment until first evidence of disease progression as per RECIST 1.1 or death from any cause.
Adverse events | Up to 4 years
  Determine toxicity, frequency, and severity of Adverse Events (CTCAE V5.0)

OTHER OUTCOMES:
Patient reported Quality Of Life (QOL) as measured by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for cancer patients (QLQ-C30) | Up to 4 years
  Examine the change in patient reported QOL over the treatment period using the questionnaire EORTC QLQ-C30
Patient reported Quality Of Life (QOL) as measured by EORTC Quality of Life questionnaire for cervical cancer patients (QLQ-CX24) | Up to 4 years
  Examine the change in patient reported QOL over the treatment period using the questionnaire EORTC QLQ-CX24

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Goh, MBBS, FRACP, Principal Investigator — Royal Brisbane & Womens Hospital

IPD SHARING:
Plan to Share IPD: No